CLINICAL TRIAL: NCT06819371
Title: Effects of Dual Task and Single Task Exercise Training on Cognitive Performance, Balance and Functionality in Patients With Type 2 Diabetes
Brief Title: Impact of Dual vs. Single Task Exercise on Cognitive Function, Balance, and Functionality in Type 2 Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Ferruh Taşpınar, Prof. Dr., Izmir Democracy University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dualtask
Record Dates: First submitted 2025-01-23; First posted 2025-02-11 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Diabetes Mellitus Type 2; Dual task; Cognitive Function; Balance
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (No Intervention): No exercise will be applied. Patients will walk 60 minutes a week for 8 weeks
- single task exercise group (Experimental): 12 participants will do balance exercises focusing on a single task for 8 weeks
  Interventions: Other: Single Task Exercise
- dual task exercise group (Experimental): 12 participants will perform a simultaneous cognitive task in addition to balance exercise for 8 weeks
  Interventions: Other: Single Task Exercise; Other: Dual Task Exercise

INTERVENTIONS:
Other: Single Task Exercise — Patients will follow the exercises in a way to focus on only one task during the exercise sessions. In the creation of the exercise programme, the principles of the exercise prescription recommended by the American Sports Medicine Association for individuals with adult Type 2 diabetes will be taken into consideration. In this context, planning will be made by considering the progression of stretching, balance and walking exercises from simple to difficult.
  Other Names: STE
  Arms: dual task exercise group; single task exercise group
Other: Dual Task Exercise — Patients enrolled in the dual-task exercise group will perform a second task during the exercise sessions along with the exercises in the single-task exercise group. This second task will be determined individually according to the level and progress of the patient.
  Other Names: DTE
  Arms: dual task exercise group

SUMMARY:
Diabetes Mellitus is defined as a carbohydrate mechanism disorder in which glucose cannot be used as an adequate energy source and is produced excessively, causing hyperglycemia. For the diagnosis of diabetes, an increase in HbA1c in the blood or a high glucose concentration in venous plasma is examined. Although there are various clinical subtypes, Type 2 diabetes constitutes 90% of the approximately 537 million diabetics worldwide. In the treatment of diabetes, there are pharmacological treatments and lifestyle changes to ensure glycemic control. The most important lifestyle change interventions are balanced calorie intake, increased physical activity and regular exercise.

The effect of exercise on complications associated with Type 2 diabetes, such as improving glycemic control, reducing inflammation and reducing cardiovascular risk, is clear and it is known that these also affect cognition.

In this context, dual-task exercises that can target both the improvement of parameters related to postural control and balance as a physical development and the development of cognitive functions are gaining importance. The aim of dual-task exercises is to direct the person's attention to another source while the first task is being performed. When the literature is examined, there are separate studies on the effects of dual-task exercises on both balance and walking performance and cognitive functions. However, the meta-analyses conducted on these studies emphasize the need for more newly designed studies. Therefore, our study aims to examine the effects of dual-task exercise training, which includes both physical and cognitive parameters, on cognitive functions, balance and functionality in individuals with type 2 diabetes. Patients who applied to the Artvin State Hospital Internal Medicine polyclinic and were diagnosed with type 2 diabetes and who meet the inclusion and exclusion criteria will be included in our study. The patients included in the study will be divided into 3 groups: dual-task exercise group, single-task exercise group and control group. Both intervention groups will be included in an exercise program with a physiotherapist 2 days a week for 8 weeks in addition to their medical treatments. The control group will be recommended walking only in addition to their medical treatment during these 8 weeks. All 3 groups will be evaluated twice, at the beginning of the study and at the end of the 8th week.

DETAILED DESCRIPTION:
Diabetes Mellitus is defined as a carbohydrate mechanism disorder in which glucose cannot be used as an adequate energy source and is overproduced, causing hyperglycemia. Diabetes is diagnosed by an increase in HbA1c in the blood or a high glucose concentration in venous plasma. Although there are various clinical subtypes, Type 2 diabetes accounts for 90% of the approximately 537 million diabetics worldwide. In the treatment of diabetes, there are pharmacological treatments and lifestyle changes to achieve glycemic control. The most important lifestyle change interventions are balanced calorie intake, increased physical activity and regular exercise.

The effect of exercise on complications associated with Type 2 diabetes, such as improving glycemic control, reducing inflammation and reducing cardiovascular risk, is clear and is known to affect cognitive functions.

Loss of postural balance is a significant problem frequently observed in patients with T2DM. Balance is defined as the individual's capacity to maintain or regulate the center of mass within the limits of balance. In this process, the integration of physiological systems including motor, sensory and dynamic control systems, vestibular, visual and proprioceptive mechanisms, muscle strength and reaction times plays a critical role. Although balance dysfunctions are generally attributed to diabetic peripheral neuropathy (DPN), balance disorders are also observed in individuals without DPN. Impaired balance function increases the risk of falling, especially in elderly T2DM patients.

However, an important problem that is frequently observed in T2DM patients but can be neglected is cognitive dysfunction. Cognitive dysfunction is a broad concept that encompasses deficiencies in various areas such as attention, memory, executive functions, language and spatial skills. Diabetes and cognitive dysfunction are chronic conditions that are frequently seen together, especially in elderly individuals, and when evaluated together, they significantly increase the risk of morbidity and mortality. Cognitive impairment can lead to serious difficulties in meeting the self-care needs of diabetic individuals and maintaining their economic and social independence. On the other hand, inadequate management of diabetes can also increase the risk of cognitive dysfunction and cause this situation to worsen.

In this context, dual-task exercises that can target both the improvement of parameters related to postural control and balance as physical development and the development of cognitive functions are gaining importance. Therefore, our study aims to examine the effects of dual-task exercise training, which includes both physical and cognitive parameters, on cognitive functions, balance and functionality in individuals with type 2 diabetes.

Patients who apply to the Artvin State Hospital Internal Medicine polyclinic and are diagnosed with type 2 diabetes and meet the inclusion and exclusion criteria will be included in our study. The patients included in the study will be divided into 3 groups: dual-task exercise group, single-task exercise group and control group.

Each of the 3 groups will be evaluated twice, at the beginning of the study and at the end of the 8th week.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with T2DM,
* Being between the ages of 40-65,
* Being able to walk independently,
* Being willing to exercise at least 2 days a week in the intervention groups as required by the research,
* Not having cooperation and communication problems,
* Not having participated in a regular exercise program in the last 6 months.

Exclusion Criteria:

* Patients who do not volunteer to participate in the study
* Patients with complications such as diabetes-related nephropathy, neuropathy, retinopathy
* Patients with orthopedic, neurological, surgical problems that prevent them from walking and exercising
* Patients with cardiac, pulmonary, or systemic diseases that prevent them from exercising
* Patients with vision problems that cannot be corrected with glasses or lenses
* Patients with hearing loss that cannot be corrected with hearing aids

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Timed get-up-and-go test (TUG) | At baseline and after 8 weeks
  It is an easy-to-administer test used to evaluate the walking speed and functional mobility of the person. At the beginning of the test, the participant is seated in a chair. With the practitioner's start command, he/she gets up from the chair and walks 3 metres to the marked point and back. Then he sits back in the chair. The time is recorded during this performance. The test is repeated 3 times and the average of the times is determined as the person's Timed get up and walk test score .
Four-step Square Test (FSST) | At baseline and after 8 weeks
  This test is a tool used to test the dynamic aspect of balance and postural control during change of direction. To perform the test, 4 equal squares are marked on the floor with a stick, stick or tape. Each of the squares is numbered from 1 to 4 and the order of the numbers is taught to the patient. The person is asked to proceed to the square where he/she takes the first step (1), the square opposite (2), the square diagonally (3) and the back side square (4) in order. Then, he/she is instructed to go back to the starting point by moving in the opposite direction and a trial is made. They are instructed not to touch the field markings when completing this cycle. The completion time of the test is measured and the best time after 3 repetitions is recorded.
Balance Error Scorring System (BESS) | At baseline and after 8 weeks
  This test is used to assess the postural control of a person on different surfaces and in different postures. For the assessment, individuals are asked to maintain the two-foot on the ground, one-foot on the ground and tandem posture positions for 20 s on both stable and unstable ground, with eyes closed. During the test, 6 situations that are accepted as errors are indicated to the individuals in advance and the test is started after they make a trial for each posture. All test steps are recorded by video recording and 20 seconds are given for each position. The person's score is calculated on the basis of the number of errors made. In the interpretation of the test, there is an inverse relationship between the number of error points and postural control.
Functional Reach Test (FRT) | At baseline and after 8 weeks
  n this test, which is used to assess dynamic balance, the participant is asked to stand sideways in front of a flat wall and extend the arm on the wall side forwards with the shoulder flexed at 90 degrees and the elbow in extension. In this position, the 3rd metacarpal joint level of the hand is marked on the wall. The person is then asked to reach as far as he/she can reach forwards without flexing the knees and without taking a step. The distance between the first marked point and the reaching point is measured with a tape measure.
Montreal Cognitive Assessment (MOCA) | At baseline and after 8 weeks
  It has an application time of approximately 10 minutes with sections including orientation ability, attention, memory, language functions, visual spatial skills and executive function processes. The score range to be obtained from the scale is between 0 and 30 and a score above 21 is considered normal.
Scoring Range | At baseline and after 8 weeks
  The test consists of two stages as forward and backward number range. For both stages, number sequences are given to the person with one second intervals. The person is asked to say the numbers in the same order for the forward range and in reverse order for the backward range. If the person cannot repeat two consecutive number sequences, the previous number sequence is recorded as the score obtained.
Stroop Test | At baseline and after 8 weeks
  The aim of the Stroop test is to evaluate the person's speed of processing information, especially simple and complex attention, inhibition ability, ability to be resistant to interference. The test to be used in our study includes 3 steps: In the first step, the person is asked to say the colours of the boxes in the form, in the second step to read the words in the form quickly, and in the last step to say the colours of the words. The time taken to complete each step is noted. The time difference between steps 2 and 3, the error made and the self-correction scores are recorded.
The Controlled Oral Word Association Test | At baseline and after 8 weeks
  In this two-stage test, both semantic and phonemic fluency are measured in order to test the person's executive function skills such as verbal fluency, mental flexibility, information processing speed, inhibition and semantic organisation. In the first stage, the person is given 1 minute and asked to produce words in a certain category (animal names). In the second stage, the person is asked to produce words starting with the letters K, A, S in 1 minute periods.

CONTACTS AND LOCATIONS:
Overall Officials: Sidrenur Aslan Kolukısa, MSc Pt, Study Director — Izmir Democracy University
Locations (1):
- Izmir Democracy University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No